CLINICAL TRIAL: NCT00733603
Title: A Single-Blinded Randomized Multi-Center Trial to Evaluate the Efficacy and Durability of Myofascial Tissue Manipulation in Women With Interstitial Cystitis/Painful Bladder Syndrome
Brief Title: Physical Therapy in Women With Interstitial Cystitis
Acronym: IC03
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ICCRN RCT3 - PT; U01DK065209 (NIH)
Record Dates: First submitted 2008-08-12; First posted 2008-08-13 (Estimated); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Interstitial Cystitis; Painful Bladder Syndrome
Keywords: Interstitial Cystitis; IC; Painful Bladder Syndrome; PBS; Bladder Pain; Pelvic Pain
MeSH Terms: conditions — Cystitis, Interstitial; Pelvic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Global Therapeutic Massage (GTM) (Sham Comparator): Non-specific somatic treatment with full-body Western massage.
  Interventions: Other: Global Therapeutic Massages (GTM)
- Myofascial Tissue Manipulation (MTM) (Active Comparator): Targeted internal and external Connective Tissue Manipulation focusing on the muscles and connective tissues of the pelvic floor, hip girdle, and abdomen.
  Interventions: Other: Myofascial Tissue Manipulation (MTM)

INTERVENTIONS:
Other: Global Therapeutic Massages (GTM) — Non-specific somatic treatment with full-body Western massage.
  Arms: Global Therapeutic Massage (GTM)
Other: Myofascial Tissue Manipulation (MTM) — Targeted internal and external Connective Tissue Manipulation focusing on the muscles and connective tissues of the pelvic floor, hip girdle, and abdomen.
  Arms: Myofascial Tissue Manipulation (MTM)

SUMMARY:
There are many different treatments that doctors recommend for patients with IC/PBS. Only a few research studies have been done to evaluate treatments given to patients. Treatment choices can be of two types: drug therapy and non-drug therapy. The two treatments used in this study will be of the non-drug therapy type. One of the treatments being used in this study is called Myofascial Tissue Manipulation. This is a kind of physical therapy that is designed to work on specific muscles and tissue layers in a particular part of the body. In this study, this treatment will focus on the areas around the pelvis and the pelvic floor. The treatment will involve the physical therapist's use of hands and fingers to target specific muscles and tissues located within your pelvis, rectum, and/or vagina (the pelvic floor) as well as muscles and layers of tissue in your abdomen and legs. The other treatment being used in this study is Global Therapeutic Massage. This treatment involves the physical therapist's use of classic Western body massage techniques on the muscles of your arms, legs, hands, neck, shoulders, back, stomach, buttocks, and feet to create an overall feeling of well being.

The purpose of this research study is to find out if Pelvic Physical Therapy is safe and effective on treating symptoms in women with interstitial cystitis as compared to a full body therapeutic massage. This study will also measure the lasting effects of the treatment up to 3 months after your last study treatment.

DETAILED DESCRIPTION:
The Urologic Pelvic Pain Syndromes (UPPS) are characterized by pelvic pain with concurrent urinary symptoms. Broadly, the UPPS comprise Interstitial Cystitis/Painful Bladder Syndrome (IC/PBS) in men and women, and Chronic Prostatitis/Chronic Pelvic Pain Syndrome (CP/CPPS) in men, although the focus of this protocol is exclusively women with IC/PBS.

Interstitial Cystitis (IC) is a debilitating bladder disorder characterized by urinary urgency, frequency, and pain. The presentation of symptoms can be quite variable among patients, suggesting that IC is a multi-factorial syndrome with several proposed etiologies, some of which may be interrelated.1 Painful Bladder Syndrome (PBS), as defined by the International Continence Society, is "the complaint of suprapubic pain related to bladder filling, accompanied by other symptoms, such as increased daytime and night-time frequency, in the absence of proven urinary infection or other obvious pathology. 2" PBS is a clinical description of disease based on the patient's symptoms and does not depend on urodynamic or cystoscopic findings. These symptoms may be related to interstitial cystitis, although diagnostic criteria are still lacking for this entity, and the relationship between PBS and interstitial cystitis is not clear. For clarity and compliance with current nomenclature, this protocol will use the term IC/PBS.

As with many chronic pain disorders, IC/PBS is poorly understood, poorly characterized, and treatment is mostly empirical and unsatisfactory. Several proposed etiologic theories include (1) increased bladder epithelial permeability, (2) activation of bladder mast cells, (3) allergic or autoimmune processes, (4) toxic substance(s) in the urine, (5) occult infection, (6) neuropathic changes, and (7) neurogenic inflammation. However, none of these mechanisms have been conclusively shown to be responsible for IC/PBS. Estimates of prevalence of the syndromes vary widely. In 1990 interstitial cystitis (IC) was thought to affect as many as 500,000 U.S. citizens, with 25% of patients under age 25.3 More recently however, using expanded definitions of PBS now exceed 10 million.4 Quality of life with IC/PBS can be worse than end stage renal disease.5 The recent pilot study of manual physical therapies for Urologic Pelvic Pain demonstrated feasibility of recruitment, and promising benefit of myofascial tissue manipulation (MTM) (ref manuscript#1). In that pilot study, 47 participants were recruited to six centers with prior expertise in MTM. Of the 47 participants, 24 were females with IC/PBS, and 23 were males -- 2 with IC/PBS and 21 with CP/CPPS. Motivated by the promising findings in that pilot study, this protocol aims to investigate whether those initial results are generalizable in an expanded phase 3 clinical trial, in which we include other therapists from other centers. However, due to the gender-specific findings of the pilot study, and the limited resources available, this protocol is focused on replicating the initial pilot study exclusively in women with IC/PBS.

Although the pain of IC/PBS is poorly understood, almost all clinicians agree that there is almost always some chronic tension and tenderness of the pelvic floor musculature present in UPPS patients,8-10 and it is possible that these myofascial abnormalities contribute significantly to the pain of IC/PBS. For example, Hetrick et al11 compared the surface EMG signals from men with CPPS to those from men without chronic pain, and found that there was greater EMG instability in men with CPPS, along with increased baseline tonicity, and instability with lowered voluntary endurance contraction amplitude.

Whether these musculoskeletal abnormalities of the abdominal wall and pelvic floor musculature found in IC/PBS sufferers represent primary or secondary phenomena remains unknown. It is possible that pelvic visceral pain leads to chronic contraction of regional skeletal musculature, leading to overuse injury and pain. It is also possible that primary pelvic myofascial problems lead to painful and weakened pelvic floor musculature, which also functions poorly to inhibit the urgency associated with bladder filling.

Our prior study of manual physical therapy suggested benefit of MTM over GTM. Translation of those office practices into the research setting was apparently successful in centers that participated in the first trial. We propose to expand the number of treating therapists to include 11 study centers, in order to determine whether the results of the first trial can be generalized, at least in the research setting. However, due to the gender-specific findings, this expanded replication study will focus exclusively on women with IC/PBS.

ELIGIBILITY:
Inclusion Criteria:

* Participant has signed and dated the appropriate Informed Consent document.
* Female participant is ≥ 18 years of age.
* Currently using an approved method of birth control, or surgically sterile, or of non-child bearing age with no menstrual period for the past year.
* Participant has a clinical diagnosis of IC/PBS in the opinion of the investigator.
* Participant with IC/PBS has reported a bladder pain/discomfort score of 3 or greater on a 0-10 Likert scale over the previous four weeks. This bladder pain/discomfort criterion must be met at each of the two baseline screening visits as reported by the participant.
* Participant with IC/PBS has reported a symptom score of abnormal urinary frequency of 3 or greater on a 0-10 Likert scale over the previous four weeks. This frequency criterion must be met at each of the two baseline screening visits, as reported by the participant.
* Participant has had symptoms of discomfort or pain in the pelvic region for at least a three (3) month period within the last six (6) months.
* Current symptoms have been present for less than 3 years. If similar symptoms were present in the past, they must have been completely resolved for at least one year prior to onset of current symptoms.
* Participant has previously undergone at least one course of therapy (other than physical therapy) for her symptoms.
* Presence of tenderness/pain to palpation found by the physician in one of the pelvic floor musculature domains during the first baseline screening visit physical examination which are confirmed by the physical therapist at screening visit 2. Presence of tenderness/pain is defined as a mild, moderate or severe finding by the physician at visit 1 and physical therapist at visit 2. The pelvic floor musculature domains are defined as: anterior or posterior levator muscles, obturator internus muscles and urogenital diaphragm (bulbospongiosus, superficial transverse perinei, ischiocavernosus, central tendon/perineal body). The assessment of tenderness/pain at Visits 1 and 2 do not need to be identical in severity or location in order for the participant to be eligible.

Exclusion Criteria:

* Participant has relevant, painful scars on lower abdominal wall that, in the opinion of the study physician or physical therapist, is unlikely to respond to physical therapy without adjuvant therapy such as injection /needling.
* A positive urine culture (defined as >100,000 CFU/ml) is exclusionary. A negative urine culture within 1 month of study enrollment is acceptable.
* Participant is unable to tolerate insertion of one or two vaginal examining fingers (e.g. vulvar allodynia), or one rectal examining finger.
* Participant had prior course of physical therapy that included manual therapy with connective tissue manipulation by physical therapist for same symptoms. Prior treatment by therapist with biofeedback, electrical stimulation, or pelvic floor exercises is not exclusionary.
* Participant has relevant neurologic disorder that affects bladder and/or neuromuscular function in the opinion of the investigator.
* Participant has active urethral or ureteral calculi, urethral diverticulum.
* Participant has a history of pelvic radiation therapy, tuberculous cystitis, bladder cancer, carcinoma in situ, or urethral cancer.
* Participant has/reports any severe debilitating or urgent concurrent medical condition.
* Participant has a potentially significant pelvic pathology or abnormalities on examination or prior imaging, including prolapse beyond the hymenal ring, pelvic mass, etc. that could cause or contribute to the clinical symptoms or require treatment.
* Participant is unlikely to be compliant due to unmanaged medical or psychological condition, including neurological, psychological or speech /language problems that will interfere with her ability to complete the study.
* Participant has an imminent change in residence or other social factors that could compromise compliance with the protocol.
* Pregnancy or refusal of medically approved/reliable birth control in women of child-bearing potential.
* Participant has pain, frequency, urgency symptoms present only during menses.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2008-06 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Proportion of responders moderately or markedly improved on a 7-point global response assessment (GRA) scale | 12 Weeks
  The GRA asked: "As compared to when you started the current study, how would you rate your overall symptoms now?" the 7 response options were markedly worse, moderately worse, slightly worse, the same, slightly improved, moderately improved and markedly improved

SECONDARY OUTCOMES:
Change in pain score | Baseline and 12 weeks
  Change from baseline to 12 weeks in a 0-10 Likert scale where higher scores indicate worse pain
Change in urgency score | Baseline and 12 weeks
  Change from baseline to 12 weeks in a 0-10 urinary urgency scale where higher scores indicate more urgency
Change in frequency score | Baseline and 12 weeks
  Change from baseline to 12 weeks in a 0-10 urinary frequency scale where higher scores indicate greater frequency

CONTACTS AND LOCATIONS:
Overall Officials: LeRoy M Nyberg, MD, PhD, Study Director — NIDDK/NIH; Mary P Fitzgerald, MD, Study Chair — Loyola University; Richard Landis, PhD, Principal Investigator — University of Pennsylvania; Robert Mayer, MD, Principal Investigator — University of Rochester; Emily Lukacz, MD, Principal Investigator — University of California, San Diego; Kenneth Peters, MD, Principal Investigator — William Beaumont Hospital, Royal Oak, MI; Toby Chai, MD, Principal Investigator — University of Maryland, College Park; Christopher Payne, MD, Principal Investigator — Stanford University; Claire Yang, MD, Principal Investigator — University of Washington; Phillip Hanno, MD, Principal Investigator — University of Pennsylvania; Karl Kreder, MD, Principal Investigator — University of Iowa; David Burks, MD, Principal Investigator — Henry Ford Hospital, Detroit; Curtis Nickel, MD, Principal Investigator — Queen's University, Ontario, Canada; Harris Foster, MD, Study Chair — Yale University
Locations (11):
- United States (10):
  - Univeristy of California San Diego, San Diego, California
  - Stanford University Medical center, Stanford, California
  - Loyola University Medical Center, Maywood, Illinois
  - University of Iowa Hospitals and Clinic, Iowa City, Iowa
  - University of Maryland, Baltimore, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - University of Rochester Medical Center, Rochester, New York
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - University of Washington, Seattle, Washington
- Queen's University, Kingston, Ontario, Canada

REFERENCES:
- [Result] FitzGerald MP, Payne CK, Lukacz ES, Yang CC, Peters KM, Chai TC, Nickel JC, Hanno PM, Kreder KJ, Burks DA, Mayer R, Kotarinos R, Fortman C, Allen TM, Fraser L, Mason-Cover M, Furey C, Odabachian L, Sanfield A, Chu J, Huestis K, Tata GE, Dugan N, Sheth H, Bewyer K, Anaeme A, Newton K, Featherstone W, Halle-Podell R, Cen L, Landis JR, Propert KJ, Foster HE Jr, Kusek JW, Nyberg LM; Interstitial Cystitis Collaborative Research Network. Randomized multicenter clinical trial of myofascial physical therapy in women with interstitial cystitis/painful bladder syndrome and pelvic floor tenderness. J Urol. 2012 Jun;187(6):2113-8. doi: 10.1016/j.juro.2012.01.123. Epub 2012 Apr 12. PMID 22503015
- [Derived] Imamura M, Scott NW, Wallace SA, Ogah JA, Ford AA, Dubos YA, Brazzelli M. Interventions for treating people with symptoms of bladder pain syndrome: a network meta-analysis. Cochrane Database Syst Rev. 2020 Jul 30;7(7):CD013325. doi: 10.1002/14651858.CD013325.pub2. PMID 32734597